CLINICAL TRIAL: NCT06390800
Title: Personalized Motor Learning in Primary Care Physiotherapy; A Prospective Formative Process Evaluation
Brief Title: Personalized Motor Learning in Primary Care Physiotherapy (TREAT)
Status: Completed | Type: Observational
Sponsor: Zuyd University of Applied Sciences (Other)
Collaborators: Fysio Bunde (Unknown); Fysio Regtop (Unknown); Fysiotherapie zesgehuchten (Unknown); Fysiotherapie Veldhoven zuyd (Unknown); Fysiotherapie ART-health (Unknown); Fysio van het Hoof (Unknown); Fysiotherapie Corine Cuijpers (Unknown); Frank Helgers (Unknown); Fysiotherapie Kemps-Rijf (Unknown); Cerfontaine&vanderLoop (Unknown); Fysiotherapie Denssana (Unknown); Maastricht Universitair Medisch Centrum (Unknown); Regieorgaan SIA (Unknown); Brunel University London (Unknown); Fontys Paramedische Hogeschool (Unknown); Kennisnetwerk CVA Nederland (Unknown); Koninklijk Nederlands Genootschap voor Fysiotherapie (KNGF) (Unknown)
Responsible Party: Sponsor
Other Study IDs: METCZ20230061
Record Dates: First submitted 2023-09-13; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Geriatric Patients; Neurological Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over the last decade many scientific articles have been published on motor learning in neurological and geriatric rehabilitation. To make the available findings comprehendible and clear for physiotherapists, a card set and website have been developed.

The aim of this prospective study is to evaluate the use and experiences of the card set and website designed to aid the physiotherapist in decision making with regards to motor learning. The following research question is central to this evaluation: How are the developed card set and website used and experienced by physiotherapists in primary care during the treatment of patients with neurological or geriatric conditions?

DETAILED DESCRIPTION:
Method: Formative process evaluation.

Over the last decade many scientific articles have been published on motor learning in neurological and geriatric rehabilitation. To make the available findings comprehendible and clear for physiotherapists, a card set and website have been developed. Participating physiotherapists will use the "card set and website" in their daily practice for a period of six months. To assess the usage and experiences of therapists, digital questionnaires will be administered prior to the intervention, at 3 months, and at 6 months, along with bi-weekly monitoring. The quantitative data from the questionnaires and monitoring will be analyzed using descriptive statistics (e.g., frequency tables, means, medians, IQR, and summary figures). Additionally, an interim evaluation will take place where solutions for the main user issues will be collectively brainstormed with the participants. Finally, a consensus meeting will be held to reach the final versions of the card set and website. The nominal group technique will be used to ensure active participation from all participants and to achieve consensus on the definitive list of modifications.

ELIGIBILITY:
Physiotherapists will be eligible for inclusion when they:

* have at least one year of working experience
* are treating neurological and/or geriatric patients
* are able to attend the preparatory training provided by the researchers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy working physiotherapist will be included for this study to help evaluate the card set and website
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Questionnaire | Six months
  A qualitative questionnaire will be filled in three times throughout the study. This questionnaire inquires participants' experience regarding the card set and website.
Monitor | Six months
  A quantitative questionnaire will be filled in biweekly. This questionnaire assesses the frequency of usage of the card set and website
Midterm evaluation | At three months into the study
  This meeting will be held to further specify and solve user problems. During this in-person session, problems that arise during the usage of the material will be discussed in depth under supervision from an experienced researcher. The meeting will be audio recorded whereafter it will be transcribed and analyzed into clusters and themes.
Consensus meeting | At six months into the study
  The goal of this meeting is to reach a final version of the card set and website based on the experiences from the process evaluation. During the in-person session, a nominal group method will ensure consensus regarding possible changes to the material and future directions the material should take e.g., more emphasis on the analogue or digital component or implementation into education. Through communal voting participants will make decisions regarding possible solutions or directions of the material. The session will be audio recorded and transcribed for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Juan Jie, PhD, Principal Investigator — Zuyd University of Applied Sciences; Guus Rothuizen, MSc, Principal Investigator — Zuyd University of Applied Sciences
Locations (1):
- Zuyd University of Applied Sciences, Heerlen, Limburg, Netherlands

REFERENCES:
- [Background] Kleynen M, Beurskens A, Olijve H, Kamphuis J, Braun S. Application of motor learning in neurorehabilitation: a framework for health-care professionals. Physiother Theory Pract. 2020 Jan;36(1):1-20. doi: 10.1080/09593985.2018.1483987. Epub 2018 Jun 19. PMID 29920128
- See also: The developed website to be evaluated in this project — http://www.motorisch-leren.nl